CLINICAL TRIAL: NCT06423846
Title: Comparison of Total Intravenous Anesthesia Versus Inhalation Anesthesia on Postoperative Liver Function in Patients With Non-Alcoholic Steatohepatitis Undergoing Laparoscopic Sleeve Gastrectomy: A Randomized Clinical Trial
Brief Title: Total Intravenous Anesthesia Versus Inhalation Anesthesia on Postoperative Liver Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ramy Mousa, Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-3-4-2024
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Laparoscopic Sleeve Gastrectomy
Keywords: Total Intravenous Anesthesia; Inhalation Anesthesia; Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: The participants were randomized into two equal groups using a computer-generated list of random numbers sealed in an opaque envelope and were randomly allocated into two groups on a scale of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total intravenous anesthesia group (Experimental): Patients in the TIVA group had anesthesia induced with propofol 2 mg/kg , fentanyl 1 ug/kg and maintained with propofol.
  Interventions: Drug: Total intravenous anesthesia group
- sevoflurane group (Experimental): general anesthesia was induced with propofol 2 mg/kg, fentanyl 1 ug/kg and then maintained with sevoflurane in air and oxygen, dexmedetomidine 1 ug/kg/hour.
  Interventions: Drug: sevoflurane group

INTERVENTIONS:
Drug: Total intravenous anesthesia group — Patients in the TIVA group had anesthesia induced with propofol 2 mg/kg , fentanyl 1 ug/kg and maintained with propofol. 200 ug/kg/min, fentanyl 0.1ug/kg/min, dexmedetomidine 1 ug/kg/hour
  Other Names: TIVA group
  Arms: total intravenous anesthesia group
Drug: sevoflurane group — For patients in the SEVO group, general anesthesia was induced with propofol 2 mg/kg, fentanyl 1 ug/kg and then maintained with sevoflurane in air and oxygen, dexmedetomidine 1 ug/kg/hour.
  Other Names: SEVO group
  Arms: sevoflurane group

SUMMARY:
The pandemic of obesity has become a serious issue of public health worldwide as the size of the obese population has almost tripled over the last four decades and continues to riseزThe epidemic of obesity has led to a significant increase in the prevalence of non-alcoholic fatty liver disease (NAFLD). NAFLD is currently the most common chronic liver disease, with an estimated global prevalence at 25-30%, rising up to 90% in morbidly obese patients

DETAILED DESCRIPTION:
Anesthesia and surgery may deteriorate liver function in patients with elevated liver enzyme levels; therefore, in these patients, choosing anaesthetics with less hepatotoxicity may be important. Halothane, which is a typical inhalational anesthetic, is known for its liver and kidney toxicity. The latest anesthetic agents, including sevoflurane and desflurane, are associated with less hepatotoxicity, although rare cases of acute liver injury have been reported with these agentsزPropofol (2,6-diisopropylphenol) is an intravenous anesthetic. Its pharmacokinetic profile makes it very suitable for total intravenous anesthesia (TIVA) and this is a widely used technique in many centers. Its use results in a rapid onset and offset with fewer side effects including postoperative nausea and vomiting, making it particularly favorable in the ambulatory setting

ELIGIBILITY:
Inclusion Criteria:

* Obese patients
* had ASA I-III
* diagnosed with non-alcoholic steatohepatitis (NASH) liver disease
* undergoing laparoscopic sleeve gastrectomy

Exclusion Criteria:

* cases wherein surgeries were performed using anesthetic methods that were not clearly identified as TIVA or INHA
* heart surgery or cesarean section, and cases of neuromuscular diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-12 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | visual analogue scale was measured at day one and day two postoperatively
  Pain was assessed by using the visual analogue scale (VAS) score for pain (0-no pain, 10-worst imaginable pain)

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  5-point Likert scale, (1=extremely dissatisfied; 5=extremely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Saleh, MD, Principal Investigator — Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed OT, Gidener T, Mara KC, Larson JJ, Therneau TM, Allen AM. Natural History of Nonalcoholic Fatty Liver Disease With Normal Body Mass Index: A Population-Based Study. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1374-1381.e6. doi: 10.1016/j.cgh.2021.07.016. Epub 2021 Jul 13. PMID 34265444